CLINICAL TRIAL: NCT02824822
Title: Genetic Markers of Cardiovascular Diseases and the Potential Role in Sudden Unexpected Death in Epilepsy.
Brief Title: Genetic Markers of Cardiovascular Disease in Epilepsy
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Virend Somers, MD, PhD, PI, Mayo Clinic
Other Study IDs: 15-002420
Record Dates: First submitted 2016-06-22; First posted 2016-07-07 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Epilepsy; Seizures; Syncope; Channelopathy; Cardiomyopathies
Keywords: Sudden Unexpected Death in Epilepsy; SUDEP; Sudden Cardiac Arrest; Sudden Cardiac Death; Sleep; Ion channel disease; Long QT syndrome; Brugada; Catecholaminergic Polymorphic Ventricular Tachycardia
MeSH Terms: conditions — Epilepsy; Seizures; Syncope; Channelopathies; Cardiomyopathies; Sudden Unexpected Death in Epilepsy; Death, Sudden, Cardiac; Long QT Syndrome; Polymorphic Catecholaminergic Ventricular Tachycardia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 50 mls of blood from a vein will be drawn at Mayo Clinic or another medical center and returned through the mail. Buccal swabs will be collected using a swab and saliva based-kit.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High SUDEP risk cohort: Patients with epilepsy who have a high SUDEP-7 risk score and/or a blood-relative with epilepsy, seizure, cardiac arrest, sudden death, drowning/near-drowning, syncope or arrhythmia.
- Low SUDEP risk cohort: Patients with epilepsy and a low SUDEP-7 score.

SUMMARY:
Epilepsy is a common condition which affects over 3 million people in the US. Patients with uncontrolled epilepsy have a lifetime risk of sudden unexpected death (SUDEP) of 35%, which is greatest in those under 40 years of age. The exact mechanisms and causes are not understood but can be due to underlying conditions which affect the heart and brain, which may lead to dangerous heart rhythms and death. Some of these conditions which affect heart and brain have an identifiable genetic cause. This study aims to identify known genetic causes of heart rhythm and sudden death related disorders in patients with epilepsy.

DETAILED DESCRIPTION:
The overall goals are to determine whether patients with epilepsy who have the highest risk of SUDEP have an underlying genetic cardiovascular disorder. The investigators are seeking patients with epilepsy who have a high risk of SUDEP identified by using a risk scoring tool called SUDEP-7 and/or have blood-relatives with a history of epilepsy, seizure, cardiac arrest, sudden death, drowning/near-drowning, syncope or heart rhythm disorder. The investigators may also include blood-relatives of patients with epilepsy and invite them to participate by providing a blood sample and/or buccal cells (from a swab or saliva) for genetic testing.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18 - 50 with a diagnosis of epilepsy or seizures, or syncope or drowning or cardiac arrest or sudden death or an abnormal ECG suggestive of an arrhythmia
* Blood-relatives (Aged 18+) of a patient with a history of epilepsy, seizure, cardiac arrest, sudden death, drowning, syncope or arrhythmia

Exclusion Criteria:

* Those who are unable to provide written consent.
* Prisoners (vulnerable population)
* Seizures secondary to ischemic events
* Traumatic brain injury resulting in seizures
* History of cranial surgery
* History of brain tumor

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Men and women diagnosed with epilepsy or seizures or unexplained syncope and blood relatives.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-05; Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Using Next Generation Whole-Exome Sequencing, determine if an underlying genetic cardiac mutation is present in refractory epilepsy patients who are at highest risk of sudden death. | 3-5 years
  SUDEP-7 is a risk profiling tool, with a score ranging from 0-12. Generally, a score greater than or equal to 3 is considered high risk. The investigators will select participants with a family history of epilepsy, seizures, cardiac arrest, sudden death, drowning, syncope or arrhythmia, as this markedly increases genetic yield.
  Next Generation Whole-Exome Sequencing will be performed with a focus on known genes implicated in sudden unexpected death syndromes (channelopathies, cardiomyopathies and aortopathies) and autonomic control. Where relevant, blood-relatives may be invited for genomic 'trio' analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Virend K. Somers, MD PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States